CLINICAL TRIAL: NCT04974541
Title: Improving Wellbeing in Ischemic Heart Disease: the Potential Efficacy of Digitally-delivered Psychological Interventions
Brief Title: Improving Wellbeing in Ischemic Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bryan Taylor, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21-002384
Record Dates: First submitted 2021-06-24; First posted 2021-07-23 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiac rehabilitation with standard psychosocial care plus Heart Health Yoga (Experimental): Subjects will participate in 12-weeks of cardiac rehabilitation with standard psychosocial care plus Heart Health Yoga
  Interventions: Other: Heart Health Yoga; Other: Psychosocial education
- Cardiac rehabilitation with standard psychosocial care (Active Comparator): Subjects will participate in 12-weeks of cardiac rehabilitation with standard psychosocial education component
  Interventions: Other: Psychosocial education

INTERVENTIONS:
Other: Heart Health Yoga — Yoga-based digital intervention
  Arms: Cardiac rehabilitation with standard psychosocial care plus Heart Health Yoga
Other: Psychosocial education — Standard psychosocial education component

SUMMARY:
The purpose of this research is to see if Heart Health Yoga (HHY) Program when added on to standard cardiac rehabilitation (CR) will improve overall wellbeing and quality of life for patients experiencing ischemic heart disease, heart problems caused by narrowed heart arteries.

DETAILED DESCRIPTION:
The overarching aim of this project is to evaluate the impact of adding a novel digitally-delivered wellbeing intervention, namely the Heart Health Yoga (HHY) program, on overall wellbeing and quality of life (QoL), cardiovascular risk markers, adherence to therapy, sleep quality, and recurrent hospitalizations amongst ischemic heart disease (IHD) patients undergoing cardiac rehabilitation (CR). This aim will be addressed through the following objectives:

Objective 1: Assess the clinical efficacy of the added digitally delivered HHY program compared to standard psychosocial intervention alone on overall wellbeing and QoL amongst IHD patients undergoing CR.

Aim 1 (Primary): To evaluate and compare the impact of the added digitally delivered HHY program versus standard psychosocial intervention alone on wellbeing and QoL, as assessed using the MacNew heart disease questionnaire, amongst IHD patients undergoing CR.

Objective 2: Assess the benefit of the added digitally delivered HHY program compared to standard psychosocial intervention alone on cardio-metabolic risk, therapy adherence, sleep quality, and recurrent hospitalization amongst IHD patients undergoing CR.

Aim 2 (Secondary): Assess and compare the impact of the added digitally delivered HHY program versus standard psychosocial intervention alone on cardio-metabolic risk (i.e. hs-CRP, AM cortisol, body weight, waist circumference, heart rate and blood pressure), therapy adherence (via weekly compliance questionnaire for HHY group, Medication Adherence Report Scale [MARS-5], Fitbit activity tracker), exercise capacity (6 minute walk test) and muscular strength (hand grip testing), sleep quality (measured using Fitbit), and recurrent hospitalizations (determined by 1 year hospital re-admission rates) amongst IHD patients undergoing CR.

Hypothesis: Amongst IHD patients undergoing CR, compared to current standard psychosocial interventions addition of a digitally delivered wellbeing technology will result in: 1) greater improvements in overall wellbeing and quality of life; 2) a more profound reduction in cardio-metabolic risk; 3) greater therapy adherence and improved sleep quality; 4) greater increase in physical activity and/or exercise capacity; and 5) reduced incidence of recurrent hospitalizations.

Innovation: There is sparse evidence available on digitally delivered psychosocial interventions for CR patients. A recent meta-analysis highlighted the feasibility and benefits of web and mobile-based delivery of cardiac rehabilitation interventions on healthy lifestyle changes, quality of life and re-hospitalizations; however, the evidence was of low-moderate quality. The authors also highlighted the limited evidence pertaining to psychological wellbeing and overall cardiovascular risk markers [23]. Yet another meta-analysis concluded that while eHealth is a feasible option for secondary prevention amongst patients with coronary artery disease, much heterogeneity remains regarding modes of delivery and outcome assessment. Only 6 out of 24 studies in this meta-analysis looked at psychosocial outcomes in addition to other traditional cardiovascular outcomes [24]. Based on the aforementioned considerations, it is clear that despite the potential clinical efficacy of well delivered psychosocial interventions on overall wellbeing, QoL, CV risk and outcomes, the direct impact of such interventions are chronically understudied. This will be the first study to assess the impact of individually delivered digital wellbeing technology namely "Heart Health Yoga (HHY)", on wellbeing and QoL improvement amongst IHD patients undergoing CR.

Approach: The Mayo Clinic CP Rehab program graduates ~200 cardiovascular disease patients per year, ~35% being post-PCI. We will recruit a convenience sample of these patients' over 12 months. Patients who consent to take part in this research will be allocated at random (1:1) to one of two groups: 1) cardiac rehabilitation plus "Heart Health Yoga (HHY)" or 2) cardiac rehabilitation with standard psychosocial education component. We will exclude those with cognitive impairment or those on antipsychotic medications. In addition to routine CR baseline assessments, baseline wellbeing and QoL will be assessed using the MacNew heart disease questionnaire. Outcome measures upon completion of CR will include changes in 1) Wellbeing/QoL scores, 2) Cardio-metabolic markers (hs-CRP, cortisol, body weight, waist circumference, BP, HR); 3) Therapy adherence (via weekly compliance questionnaire for HHY group, Medication Adherence Report Scale [MARS-5], Fitbit step tracker), exercise capacity (measured by 6 min walk distance) and muscular strength (measured by hand grip testing), 4) Sleep quality (measured using Fitbit) & 4) Recurrent hospitalizations at 1 year

Methods:

This is a prospective single blind randomized pilot study comparing the effects of digitally delivered HHY program vs. standard psychosocial intervention on wellbeing/QoL, cardio-metabolic risk markers, therapy adherence and recurrent hospitalizations amongst IHD patients undergoing CP rehab. Eligible participants will be recruited at their first CR visit with prospective enrollment.

Recruitment:

Patients will be recruited for the study at the time of their first visit to cardiac rehabilitation. Cardiac rehabilitation staff will offer patients the option to participate in the study and obtain consent.

Participants will need to consent to blood draws before and after the study.

Enrollment:

Interested participants will be scheduled for an initial appointment to confirm eligibility criteria, obtain consent, randomization and baseline testing Visit 1. Randomization will be done stratified on Charlson Comorbidity Index (CCI) categories (mild = CCI 1-2; moderate = CCI 3-4; severe = CCI 5 or more). To ensure near balance in the number of patients in each study arm throughout the trial, we will used blocked randomization within each CCI category randomization patients to either HHY or standard of care in a 1:1 fashion with random block sizes of 2 or 4 patients. Investigators and statistician will be blinded to participant groups until after study completion and analysis of the primary endpoint.

Consent: Participants must sign the informed consent form prior to being enrolled in the study.

Assignment: Participants will be assigned to one of the two CR groups (online HHY intervention + Standard psychosocial intervention or standard psychosocial intervention only control group).

* The HHY + Standard psychosocial care group participants will complete 6 online modules (12-25 minutes in length) sequentially on their own time between weeks 3-5. The length of time to perform all the recommended Hatha Yoga practices daily will be less than 30 minutes. For the 12-week duration of the study, Hatha Yoga Practices will be completed at least once daily. It is recommended for the participants to perform guided meditation sessions at least twice weekly. There will be 2 online group sessions available to participants for guided practice sessions. These will be timed between weeks 6-7.
* The control group is the standard psychosocial care group who will receive standard brief education/advice on psychosocial wellbeing and stress reduction.

Baseline testing Visit 1: Once consented, subjects will undergo a baseline assessment.

Baseline testing will be performed ~1-2 weeks prior to the start of digital HHY training. Baseline data collection will include height, weight, waist and hip circumference, 6 minute walk test distance, overnight fasting blood draw (cardio-metabolic biomarkers), resting blood pressure and heart rate, hand grip testing and questionnaires (Table 1). Most of the study activities will occur in CR.

Baseline questionnaires will include- MacNew Heart Disease questionnaire, Medication adherence Report Scale [MARS-5], Brief Resilience Scale and Adverse Childhood Experience questionaire. Questionnaires will be completed electronically (i.e. REDCap) or on paper. Paper data will be securely stored with locked access only accessible by relevant study personnel.

This study will utilize a commercially available wearable device (i.e. Fitbit Inspire 2) along with the research platform Fitabase to obtain sleep and activity data for 2 months on the participants. Fitbit will be mailed to participants and they will be asked to wear device as often as they can during the observation period. The participants will be able to control the Fibit.com user account (uses their own email/password) associated with the Fitbit device. They will be asked to authorize the Fitabase system via an email to access their Fitbit data and make it available for download for analysis. As appreciation for their participation, participants may keep the Fitbit device for personal use after the study period. Data will be collected via Fitabase research platform which is secure (https://www.fitabase.com/resources/knowledge-base/working-with-the-irb/). Data will be examined for objective sleep and activity parameters.

Weekly compliance questionnaires will be sent to the HHY intervention group starting week 3, to assess compliance with practices.

Visit 2 at 6 weeks:

Data collection will include height, weight, waist and hip circumference, resting blood pressure and heart rate, hand grip testing, and 6-minute walk test distance and parameters. Questionnaires will be completed (MacNew Heart Disease questionnaire, Medication adherence Report Scale [MARS-5],).

Visit 3 at 8 weeks:

Post CR testing will be performed within 1 week following the final CR session. Visit 3 data collection will include height, weight, waist and hip circumference, 6-minute walk test distance and parameters, resting blood pressure and heart rate and hand grip testing.

Questionnaires will be completed (MacNew Heart Disease questionnaire, Medication adherence Report Scale [MARS-5]).

Visit 4 at 12 weeks:

Visit 4 data collection will include height, weight, waist and hip circumference, temperature, 6-minute walk test distance and parameters, overnight fasting blood draw (cardio-metabolic markers), resting blood pressure and heart rate and hand grip testing.

Questionnaires will be completed (MacNew Heart Disease questionnaire, Medication adherence Report Scale [MARS-5]).

Other Follow-up If subjects are not able to complete the questionnaires at the visit, we can send them postage paid return envelope, follow-up by e-mail or be telephone in attempt to receive missing data.

Subjects may be contacted by telephone to remind them of their follow-up appointments, or to troubleshoot the devices, or to remind them to follow the HHY program.

Remuneration Subjects will not receive any remuneration for participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-65 years of age.
* Willing and able to provide informed consent.
* Have a computer and smartphone for access to study videos and online questionnaires, and willing and able to download Fitbit app.

Exclusion Criteria:

* Unable to provide informed consent.
* Orthopedic injury/limitation or any other contraindications to exercise.
* Known active psychiatric conditions including bipolar disorder, schizophrenia, mania, obsessive compulsive disorder.
* Active treatment with antipsychotic medications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Change in health-related quality of life | Baseline, 6 weeks
  Measured in arbitrary units using the MacNew heart disease questionnaire. The MacNew heart disease measures health-related quality of life questionnaire using a global score.

SECONDARY OUTCOMES:
6 minute walk test distance measured in meters | Baseline, 6 weeks, 8 weeks, 12 weeks
  Distance a patient can walk during a 6 min test
High sensitivity C-Reactive Protein (CRP) | Baseline, 12 weeks
  Cardiometabolic risk using high sensitivity CRP measured in mg/L
AM cortisol | Baseline, 12 weeks
  Cardiometabolic risk using AM cortisol in mcg/dL
Height | Baseline, 6 weeks, 8 weeks, 12 weeks
  Measured in centimeters (cm)
Weight | Baseline, 6 weeks, 8 weeks, 12 weeks
  Measured in kilograms (kg)
Waist circumference | Baseline, 6 weeks, 8 weeks, 12 weeks
  Measured in centimeters (cm)
Blood pressure | Baseline, 6 weeks, 8 weeks, 12 weeks
  Measured in mmHg
Heart rate | Baseline, 6 weeks, 8 weeks, 12 weeks
  Measured in beats per minute

CONTACTS AND LOCATIONS:
Overall Officials: Bryan J Taylor, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials